CLINICAL TRIAL: NCT05470296
Title: It's Native: Nudging Towards Healthy Ways in Southeastern American Indian Country
Brief Title: It's Native: Nudging Healthy Ways
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was disrupted by the COVID-19 pandemic and there it was not possible to meet study goals within the required timeframe.
Sponsor: University of Southern Mississippi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-880
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Diet, Healthy; Physical Activity
Keywords: Native American; nutrition; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Pre-/post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Move & Eat 2 Live (Other): 12, 1-hour sessions with an education and motivational component and focused on nutrition, physical activity and healthy weight.
  Interventions: Behavioral: Move & Eat 2 Live

INTERVENTIONS:
Behavioral: Move & Eat 2 Live — American Indians suffer disproportionately from several chronic diseases that may be prevented with healthier modifiable factors. Nutrition, physical activity and a healthy weight are key factors that may prevent and reduce risk of disease incidence. The major goals of this project are to develop a culturally adapted intervention that addresses barriers and uses positive cultural values as guiding principles for behavior changes to enhance program retention and improve behaviors. This project will pilot a 12-week standard lifestyle intervention in American Indians.
  Other Names: ME2L

SUMMARY:
Native Americans suffer disproportionately from chronic diseases that may be prevented by achieving a healthy diet, physical activity and weight. For this pilot study, the aim is to examine the effectiveness and feasibility of a standard lifestyle management program implemented in community based settings among Native Americans.

DETAILED DESCRIPTION:
A pilot study will be implemented to establish comparison data for the delivery of a standard lifestyle management program among Southeastern Native Americans. The program addresses the physical and intellectual domains. The ultimate goal will be to use focus group data and this pilot pre-post clinical trial to inform further cultural and social adaptations that could advance the effectiveness of lifestyle management programs in Southeastern Native Americans.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant and more than 6 months postpartum
* Without complicated disease (ie. renal failure, cancer)
* Identify as Native American
* Resident of study area
* Adults 18-50 years

Exclusion Criteria:

* Pregnant or within 6 months postpartum
* Complicated diseases states that are contraindications for the program goals
* Not Native American
* Not permanent resident of study area
* Less than 18 years of age or older than 50 years of age

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Added Sugar Intake | Change from Baseline Added Sugar Intake at 3 months
  Scale from NHANES Dietary Screener Questionnaire with higher scores meaning worse outcome
Red and Processed Meat Consumption | Change from Baseline Red and Processed Meat Intake at 3 months
  Scale from NHANES Dietary Screener Questionnaire with higher scores meaning worse outcome

SECONDARY OUTCOMES:
Physical Activity | Change from Baseline Physical Activity at 3 months
  Metabolic Equivalent of Task (MET Minutes) scale from the International Physical Activity Questionnaire with higher scores indicating better outcome
Body Mass Index | Change from Baseline Body Mass Index at 3 months
  ratio of weight (kg) to height (m2)

OTHER OUTCOMES:
Number of Participants who attend each session | up to 12 weeks
  Calculated Attendance Rate of all 12 sessions
Retention | at 12 weeks
  Percent of sample that completed the program at 12 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No